CLINICAL TRIAL: NCT02573168
Title: A Three-arm, Parallel Group, Multicentre, Double-blind, Randomized Controlled Trial Evaluating the Impact of GeneSight Psychotropic and Enhanced-GeneSight Psychotropic, on Change in Weight Following Antipsychotic Treatment in Patients Suffering From Disorders Indicated for Antipsychotic Utilization
Brief Title: Pharmacogenomic Decision Support With GeneSight Psychotropic to Guide the Treatment With Antipsychotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Programs for Assessment of Technology in Health Research Institute (Other); Centre for Addiction and Mental Health (Other); Genome Canada (Other); AssureRx Canada Ltd (Other); Assurex Health Inc. (Industry); Mars Excellence in Clinical Innovation and Technology Evaluation (Other)
Responsible Party: Principal Investigator, Jean-Eric Tarride, PI, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EXCITE-013304-ARX1010.PTL
Record Dates: First submitted 2015-10-08; First posted 2015-10-09 (Estimated); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Pharmacogenomic; Pharmacogenomic Testing; Pharmacogenomics; Genetic Testing; Genetics; GeneSight; Enhanced GeneSight; Psychotropic
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GeneSight Psychotropic (GEN) (Experimental): The GeneSight Psychotropic (GEN) product is a pharmacogenomic decision support tool that helps clinicians to make informed, evidence-based decisions about proper drug selection. More specifically, patients are tested for clinically important genetic variants of multiple pharmacokinetic and pharmacodynamic genes that affect a patient's ability to metabolize, tolerate or respond to medications.
  Interventions: Genetic: GeneSight Psychotropic (GEN)
- Enhanced-GeneSight Psychotropic (E-GEN) (Experimental): The current GEN test lacks predictive genes for antipsychotic-induced weight gain (AIWG), a major complication of antipsychotic drug use. Therefore, the Enhanced-GeneSight Psychotropic (E-GEN), which is an enhanced version of the GEN test, was developed by incorporating 6 new genes (represented by 7 SNPs) that are predictive for AIWG, to those used in the GEN algorithm. An increasing risk level associated with AIWG is estimated by an increasing number of risk genotypes that a given patient possesses among the 7 SNPs.
  Interventions: Genetic: Enhanced-GeneSight Psychotropic (E-GEN)
- Treatment as Usual (TAU) (Active Comparator): The comparator chosen for this study provides a "real world" comparison of standard of care for patients who receive no pharmacogenomics guidance.
  Patients randomized to the TAU arm will also have their DNA collected and a pharmacogenomic-based interpretive report will be generated using GEN testing. However, this report will not be shared with the treating clinicians until completion at 12 months of the study. Therefore, patients in this arm will receive clinical treatment as usual, without the use or knowledge of genotyping results by their treating clinicians.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Genetic: GeneSight Psychotropic (GEN) — Patient DNA will be collected for all subjects and measured for variations in drug target genes and in drug metabolizing genes.Recommendations for optimal choices and dose adjustments for the 33 most commonly prescribed antidepressant and antipsychotic medications will be provided to subjects randomized to the GEN arm. This pharmacogenomic-based interpretive report will be provided to treating clinicians of patients in the GEN arm of the study, allowing clinicians to use the report to support their treatment decisions.
  Arms: GeneSight Psychotropic (GEN)
Genetic: Enhanced-GeneSight Psychotropic (E-GEN) — The E-GEN test incorporates into the existing GEN product new markers that are predictive of side effect of antipsychotic-induced weight gain (AIWG). The pharmacogenomic-based interpretive report from E-GEN will be provided to treating clinicians of patients in the E-GEN arm of the study, allowing clinicians to use the report to support their treatment decisions.
  Arms: Enhanced-GeneSight Psychotropic (E-GEN)
Other: Treatment as Usual (TAU) — Subjects randomized to the TAU arm will also require collection of patient DNA. A pharmacogenomic-based interpretive report will be generated from GEN, however, this report is not provided to the treating clinician until completion of the study.
  Arms: Treatment as Usual (TAU)

SUMMARY:
Antipsychotics are approved to treat several conditions, including Schizophrenia, Schizoaffective Disorder, Bipolar Disorder, and Major Depressive Disorder among others. The typical and atypical antipsychotics, derive their therapeutic benefit predominantly from the antagonism of dopamine D2 and 5-HT2A receptors. Many of these compounds are associated with common and significant adverse effects (e.g. weight gain, extrapyramidal symptoms, hyperprolactinemia, sexual dysfunction, and cardiac effects) which negatively impact on adherence. Today, antipsychotic induced weight gain (AIWG) is a leading cause for antipsychotic discontinuation. Importantly as well, approximately 20-30% of all patients with schizophrenia do not respond adequately to an initial antipsychotic trial, and strikingly, 83% of those who go on to a second antipsychotic trial do not meet criteria for response.

To-date, no RCT has been conducted to evaluate the outcomes in patients taking antipsychotics following the use of pharmacogenomic guidance of treatment selections. Therefore, the rationale for this trial is to utilize a double-blinded RCT design to evaluate and compare the clinical outcomes in participants treated with the benefit of GEN and E-GEN testing. Furthermore, this trial also intends to develop an evidence- based case for the value of GEN and E-GEN to Canadian health-care payers.

DETAILED DESCRIPTION:
The primary objective for this study is to validate the clinical utility of the new Centre for Addiction in Mental Health (CAMH) antipsychotic induced weight gain (AIWG) markers and demonstrate the superior predictive capabilities of E-GEN as compared to GEN/TAU.

The second primary objective of this study is to compare the efficacy of GEN to treatment as usual (TAU) in improving response to psychotropic treatment in the subset of patients suffering from schizophrenia/schizoaffective disorder.

This study is designed as a three-arm multi-centre, double-blind (participants and raters), randomized controlled trial to compare the clinical and economic outcomes of GEN, E-GEN and TAU for patients suffering from psychiatric disorders indicated for antipsychotic utilization. Participants will be randomized in a 1:1:1 ratio to each of the three treatment arms. Recruitment will be 36-months and follow-up 12 months.

Subjects will complete short diagnostic interviews specific to their clinical diagnosis, basic metabolic measures (eg. blood pressure, weight), and provide buccal swab samples for genetic analysis (the unanalyzed buccal swabs and associated DNA will be biobanked). During the first visit, blood and urine samples will be required for laboratory panel screening and blood biobanking. Subjects will be monitored over a one year period and clinical measures and healthcare resource utilization will be obtained. Treating clinicians in the GEN and E-GEN arms will receive an easy to implement report providing pharmacogenomic guidance for prescribing psychotropic medications to their patients.

The study will recruit participants from 3 sites, stratified into 2 clusters. Chatham-Kent and Ontario Shores will form one of the stratified clusters. CAMH will constitute the second stratified cluster. The sample size required for this study was calculated for a large effect size (Cohen's d = 0.8) for weight change between treatment groups (GEN and E-GEN) and TAU. Sample size calculations are based on the weight gain differences observed between carriers and non-carriers of genetic risk markers in the CAMH discovery studies (18, 19, 20, 21, 22, 23). Assuming intraclass coefficient between clusters of 20%, statistical power of 80%, an alpha level of 0.05, and an expected drop-out rate of 28.3% by Week 12, a total of 90 participants (i.e., 30 per treatment arm) are required to detect the same effect in this study. Sample size calculations were determined using G*Power (version 3.1.9.2, Germany).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. Suffer from schizophrenia, schizoaffective disorder, schizophreniform disorder, psychosis not otherwise specified, bipolar disorder (I, II, NOS) or major depressive disorder meeting Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria;
3. Have moderate to severe psychiatric symptoms;
4. Intending to switch to, or start a new antipsychotic medication;:
5. Be capable and willing to provide written informed consent to participate in this study;
6. Agree to abide by the study protocol and its restrictions and be able to complete all aspects of the study, including all visits and tests.

Exclusion Criteria:

1. Patients posing a serious suicidal risk and/or violence as judged by the investigator;
2. Patients with a current Axis I diagnosis of:

   * Delirium
   * Dementia
   * Amnestic and other cognitive disorder;
3. Patients who are on restricted diets (e.g., diabetes), who have an eating restriction disorder (e.g., bulimia, anorexia), or who are undergoing weight-reducing interventions (e.g. metformin, or structured diet program).
4. Patients with a history of hypothyroidism unless taking a stable dose of thyroid medication and asymptomatic or euthyroid for 6 months;
5. Patients who meet DSM-IV-TR criteria for any significant current substance dependence;
6. Patients with:

   * hepatic insufficiency (three times the upper limit of normal (ULN) for aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT)); liver transplant recipient; cirrhosis of the liver;
   * malignancy (except basal cell carcinoma) and/or chemotherapy within 1 year prior to screening; malignancy more than 1 year prior to screening must have been local and without metastasis and/or recurrence, and if treated with chemotherapy, without nervous system complications;
   * significant unstable medical condition or life threatening disease with anticipated survival of less than 6 months;
   * need for therapies that may obscure the results of treatment and/or of the study
7. Participation in another clinical trial within 30 days of the screening visit;
8. Anticipated inability to attend scheduled study visits;
9. Patients who in the judgment of the Investigator may be unreliable or uncooperative with the evaluation procedure outlined in this protocol;
10. Patients with a history of prior pharmacogenomic testing;
11. Any change in psychotropic medication (including change in dosage) between screening and baseline;
12. Patients who are known to be pregnant or lactating;
13. Patients with a history of gastric bypass surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Change in patients' weight and waist-to-hip ratio | From baseline to week 12
  Mean change in patients' weight and waist-to-hip ratio from baseline and week 12 of the study
Change in schizophrenic symptoms as assessed by the Positive and Negative Syndrome | From baseline to Week 12
  Mean change in the PANSS score from baseline to Week 12 of the study

SECONDARY OUTCOMES:
Time between baseline and discontinuation of treatment for any cause | Baseline, Weeks 8 and 12, Months 6 and 12
Change in severity of illness as assessed by the Clinical Global Impression of Severity (CGI-S) | Baseline, Week 12, Months 6 and 12
Change in global improvement as assessed by Clinical Global Impression of Improvement (CGI-I) | Week 12, Months 6 and 12
Change in global therapeutic benefit and global severity of side effects as assessed by Clinical Global Impression Efficacy Index (CGI-EI) | Week 12, Months 6 and 12
Changes to initial prescribing based on availability of pharmacogenomic data | Screening and Baseline
Response rates to psychotropic medication | Baseline, Weeks 8 and 12, Months 6 and 12
  A responder is defined as a participant with 20% decrease in PANSS score from baseline.
Time to response | Baseline, Weeks 8 and 12, Months 6 and 12
Change in psychotropic medication side effects as assessed by the Udvalg for Kliniske Undersogeler (UKU) Side Effect Rating Scale | Baseline, Weeks 8 and 12, Months 6 and 12
Change in severity of dyskinesias as assessed by the Abnormal Involuntary Movement Scale (AIMS) | Baseline and Month 12
Change in health related quality of life as assessed by the EuroQol (EQ-5D-5L) | Baseline, Week 12, Months 6 and 12
Change in health related quality of life as assessed by the Short Form (36) Health Survey (SF-36) | Baseline, Week 12, Months 6 and 12
Pharmacogenetics in Psychiatry Follow-Up Questionnaire (PIP-FQ) | Baseline, when prescription changes are made (expected average of every 4 weeks), Months 6 and 12
  The PIPFQ is a questionnaire developed by CAMH to evaluate each physician's attitude and experience to pharmacogenomic testing. Information is solicited from the physician on three different domains: the processing of the physician's last referral, the contact and outcome of the physician's patient, and the physician's perspective on the future of genetic studies in psychiatric drug treatment.
Healthcare resource utilization (Composite measure of healthcare costs): physician visits, hospital utilization, emergency department visits, medication use, and laboratory tests | Baseline, Weeks 8 and 12, Months 6 and 12
Productivity losses (measured as economic costs) | Baseline, Weeks 8 and 12, Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Eric Tarride, PhD, Study Chair — St.Joseph's Healthcare, Hamilton/Mcmaster University; James L Kennedy, MD, Principal Investigator — Centre for Addiction and Mental Health; Bryan Dechairo, PhD, Principal Investigator — Assurex Health Inc.
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada